CLINICAL TRIAL: NCT01911013
Title: A Study of Korean Society of Spine Surgery on the Outcomes of Anterior Cervical Discectomy and Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Society of Spine Surgery (Unknown)
Responsible Party: Principal Investigator, Jin S. Yeom, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSSS-001
Record Dates: First submitted 2013-07-21; First posted 2013-07-30 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Radiculopathy, Cervical; Myelopathy
Keywords: degenerative cervical disease; anterior cervical discectomy and fusion; plate and cage; cage alone
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases | interventions — Gene Fusion; Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cage and Plate (Active Comparator): anterior cervical discectomy and fusion surgery at one segment is performed using cervical cage and plate system
  Interventions: Procedure: anterior cervical discectomy and fusion; Device: Cage and Plate
- Cage alone (Experimental): anterior cervical discectomy and fusion surgery at one segment is performed using only cervical cage without plate
  Interventions: Procedure: anterior cervical discectomy and fusion; Device: Cage alone

INTERVENTIONS:
Procedure: anterior cervical discectomy and fusion — anterior cervical discectomy and fusion with anterior plating or not
Device: Cage and Plate — anterior cervical discectomy and fusion is performed using cervical cage and plate
  Arms: Cage and Plate
Device: Cage alone — anterior cervical discectomy and fusion is performed using cage alone with plate.
  Arms: Cage alone

SUMMARY:
The purpose of this study is firstly to determine the efficacy of cervical plate for anterior cervical discectomy and fusion using cervical cage, and secondly to investigate the determining factors for surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* degenerative cervical disease
* radiculopathy or myelopathy refractory to conservative treatment
* be scheduled to undergo one segment anterior cervical discectomy and fusion
* age is more than 19 years old
* all requirements of preoperative image studies are satisfied

Exclusion Criteria:

* previous neck surgery or radiation treatments at neck area
* fusion at adjacent segments
* two segment fusion is expected
* C2-3 or C7-T1
* high risk for additional cervical surgery within one year
* ossification of posterior longitudinal ligaments, trauma, infection, tumor, congenital or developmental disease
* inadequate radiological images
* patient is not expected to be observed at long term follow-up (foreigner, international student)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cervical fusion status | five year after surgery
  Cervical fusion rates (%) is compared using CT and flexion/extension X-ray between two groups. For statistical analysis, Chi-Square test is used.

SECONDARY OUTCOMES:
predisposing factor of non-union | one year after surgery
  Using logistic regression analysis, odds ratio of each variable is calculated for non-union after anterior cervical discectomy and fusion.
risk factors of dysphagia | one year after surgery
  a specific questionnaire is used for assessment for dysphagia after anterior cervical discectomy and fusion. For comparison of dysphagia rates(%) between two group, Chi-square analysis is used. Furthermore, odds ratio of each variable for dysphagia is calculated for logistic regression analysis.
risk factors of dysphonia | one year after surgery
  a specific questionnaire is used for assessment for dysphonia after anterior cervical discectomy and fusion. For comparison of dysphonia rates(%) between two group, Chi-square analysis is used. Furthermore, odds ratio of each variable for dysphonia is calculated for logistic regression analysis.
factors for quality of life | one years after operation
  Firstly, total cost is calculated for each case. European Quality of Life-5 Dimensions is also used for assessment of quality of life after operation. Between two groups, quality of life per cost is evaluated.
risk factors for adjacent segment degeneration | five year after surgery
  The rates (%) of radiological and clinical adjacent segment degeneration is evaluated using X-ray and clinical evaluation in both groups. For statistical analysis, Chi-Square test is used for comparison of rates (%) for adjacent segment degeneration. Furthermore, logistic regression test is also used for calculating odds ratio for adjacent segment degeneration
correlation between osteoporosis and fusion | one year after surgery
  The rates (%) of fusion is evaluated in relation to osteoporosis. For statistical analysis, Chi-Square test is used for comparison between osteoporosis group and non-osteoporosis group.
relation between brace wearing and fusion | one year after surgery
  The rates (%) of fusion is evaluated using X-ray and CT scan according to kinds of brace in both groups. For statistical analysis, Chi-Square test is used for comparison of fusion rates (%).
surgical outcomes for combined uncinectomy | one year after surgery
  In relation with uncinectomy, the clinical outcomes (VAS, NDI) and radiological outcome (fusion rates(%)) is compared using t-test and Chi-square test.
change of neck motion after surgery | one year after surgery
  Serial changes of whole cervical neck motion (degree) is evaluated and compared between pre- and post-operative states. statistical significance is evaluated using one-way ANOVA or paired t test.
neuropathy after anterior cervical discectomy and fusion surgery | one year after surgery
  The occurrence rates(%) of neuropathic pain is evaluated using a specific questionnaires. Several factors to be associated with neuropathic pain is evaluated using logistic regression analysis.
relation between the method of bone graft and fusion | one year after surgery
  The rates (%) of fusion is evaluated using X-ray and CT scan according to methods of bone graft in both groups. For statistical analysis, Chi-Square test is used for comparison of fusion rates(%) in relation to the bone graft method.
analysis of complication rates after anterior cervical discectomy and fusion surgery | one year after surgery
  After anterior cervical discectomy and fusion, complication rates (%) was evaluated, and this is compared between two groups. Further, factors to be associated with complication rates is assessed using Chi-square test
The correlation between existence of co-morbidity and surgical outcome | one year after surgery
  The clinical and radiological outcomes is evaluated using VAS, NDI, and X-ray in relation with existence of coexistence. T-test and Chi-square test are used for statistical analysis for comparison between co-morbidity group and non-co-morbidity group.
The correlation analysis between smoking history and surgical outcome (fusion rates, improvement of pain and disability) | one year after surgery
  The surgical outcomes such as fusion rates(%), VAS, and NDI score were evaluated in relation with smoking history. For analysis, Chi-square and t-test are used for comparison between smoking group and non-smoking group.

CONTACTS AND LOCATIONS:
Overall Officials: Jin S. Yeom, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (31):
- South Korea (31):
  - National Health Insurance Service Ilsan Hospital, Ilsan, Gyounggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Dongan, Gyounggido
  - Hallym University Hospital, Dongan, Gyounggido
  - Inje University Ilsan Paik Hospital, Ilsan, Gyounggido
  - Bundang Jesaeng Hospital, Seongnam, Gyounggido
  - Dongguk University Ilsan Hospital, Ilsan, Gyounggi
  - CHA Bundang Medical Center, CHA university, Seongnam, Gyoungido
  - Pusan National University Yangsan Hospital, Yangsan, Gyoungnam
  - Wonkwang University School of Medicine & Hospital, Iksan, Jeollabuk-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Pohang Semyung Christianity Hospital, Pohang, Kyoungpook
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - The Catholic University of Korea Daejeon ST. Mary's hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Inha University Hospital, Incheon
  - The Catholic University of Korea, Incheon St. Mary's hospital, Incheon
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Chung-Ang University Hospital, Seoul
  - Gangnam severance hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - National Police Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - VHS Medical Center, Seoul